CLINICAL TRIAL: NCT03264651
Title: A Single-Centre Pilot Trial Investigating the Efficacy and Safety of Enobosarm and Anastrozole in Pre-menopausal Women With High Mammographic Breast Density
Brief Title: Enobosarm and Anastrozole in Pre-menopausal Women With High Mammographic Breast Density
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Havah Therapeutics Pty Ltd (Industry)
Collaborators: GTx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH02ST1
Record Dates: First submitted 2017-08-14; First posted 2017-08-29 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-02

CONDITIONS: Mammographic Density
Keywords: Selective androgen receptor modulator; Aromatase inhibitor
MeSH Terms: interventions — ostarine; Anastrozole

STUDY DESIGN:
Intervention Model Description: A single armed group of premenopausal women receiving open labeled medication
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- oral enobosarm and anastrozole (Experimental): 9 mg of oral enbosarm and 1 mg of anastrozole daily
  Interventions: Drug: enobosarm

INTERVENTIONS:
Drug: enobosarm — Oral combination therapy of enobosarm and anastrozole
  Other Names: anastrozole

SUMMARY:
To evaluate the impact of a selective androgen receptor modulator combined with an aromatase inhibitor in reducing high mammographic breast density.

DETAILED DESCRIPTION:
High mammographic breast density is a well recognized risk factor for the development of breast cancer and the masking of malignancy within the breast. Previous chemoprevention studies have revealed that only tamoxifen is efficacious in premenopausal women in the reduction of breast cancer. In order for this to occur mammographic density has to be reduced. Unfortunately the side effect profile of tamoxifen is such that not many women are taking up this therapeutic intervention. This trial is trying to establish a combination therapy to reduce mammographic breast density.

This phase 1 pilot study is combining oral enobosarm, a selective androgen receptor modulator, and oral anastrozole, an aromatase inhibitor, to study the impact of this combination treatment on mammographic breast density and breast elasticity. Safety and tolerability we also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Pre-menopausal levels of FSH/LH/E2 (follicle stimulating hormone, luteinizing hormone, oestrogen) according to the definition of "pre-menopausal range" for the laboratory involved
* Have a Volpara Density volumetric breast density of >15.5% (combined average both breasts)
* Breast pain in the previous month of equal to or greater than 40mm on a 100mm visual analogue pain scale
* WBC ≥ 3.0 x 109/L, granulocytes ≥ 1.5 X 109/L and platelets ≥ 100 x 109/L.
* AST/SGOT or ALT/SGPT ≤ 3 times ULN
* eGFR> 60 ml/min/1.73m2
* Negative pregnancy test in women of childbearing potential (premenopausal or less than 12 months of amenorrhea post-menopause, and who have not undergone surgical sterilization), no more than 7 days before the first dose of study treatment;
* For women of childbearing potential who are sexually active, agreement to use a highly effective, non-hormonal form of contraception during and for at least 6 months after completion of study treatment; OR, a fertile male partner willing and able to use effective non-hormonal means of contraception (barrier method of contraception in conjunction with spermicidal jelly, or surgical sterilization) during and for at least 6 months after completion of study treatment;

Exclusion Criteria:

* Presence of breast cancer
* Diabetes mellitus or glucose intolerance defined as a fasting glucose >6mmol/l
* Previous or concomitant other (non-breast cancer) malignancy within the previous 5 years (other than skin cancer)
* History of coronary artery disease
* Systemic hormonal contraception
* Risk of transmitting Human Immunodeficiency Virus or viral hepatitis via infected blood
* Known hypersensitivity to any component of testosterone
* Unable to comply with study requirements
* Prolonged systemic corticosteroid treatment
* Any investigational drugs
* Systemic hormone replacement therapy
* Pregnant or lactating women
* Known liver disease
* Current warfarin usage

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Mammographic breast density | 12 months
  Volumetric analysis of fibroglandular density change on mammography utilizing Volpara software
Breast tissue elasticity | 1 month
  Evaluation of breast elasticity change by direct shear wave ultrasonic measurement
Breast tissue elasticity | 3 months
  Evaluation of breast elasticity change by direct shear wave ultrasonic measurement
Breast tissue elasticity | 6 months
  Evaluation of breast elasticity change by direct shear wave ultrasonic measurement

SECONDARY OUTCOMES:
Breast pain scale | 1 month, 3 months, 12 months
  Breast pain measured on a 100 mm visual analog scale
Serum gonadotropin levels | 1 month, 3 months, 12 months
  serum follicular stimulating hormone and luteinizing hormone levels
Menopausal symptoms | 3 months, 12 months
  Menopause symptoms as recorded on a menopause symptoms scale

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N Birrell, MD PhD, Principal Investigator — Havah Therapeutics Pty Ltd
Locations (1):
- Wellend Health, Toorak Gardens, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No